CLINICAL TRIAL: NCT00056849
Title: Genetic Determinants of Ankylosing Spondylitis Severity - Cross Sectional Study
Brief Title: Genetic Determinants of Ankylosing Spondylitis Severity
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030130; 03-AR-0130
Record Dates: First submitted 2003-03-25; First posted 2003-03-25 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 1920-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Arthritis; Spondyloarthropathy; Spine; Hereditary; Disability; Ankylosing Spondylitis; AS; Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis; Spondylarthropathies; Spondylarthritis

SUMMARY:
This study will explore how genes-units of heredity-may influence the severity of ankylosing spondylitis. It will examine whether some genes may cause people with ankylosing spondylitis to have more rapid fusion of the bones of the spine, more difficulty performing daily activities, or be more likely to need joint surgery.

Patients who developed ankylosing spondylitis after age 16 and have had the disease for 20 years or more may be eligible for this study. The onset of disease is dated to the first appearance of symptoms of inflammatory low back pain or restricted spinal motion. Patients with a spondyloarthropathy other than AS may not enroll.

Participants will complete a brief medical history and physical exam. They will fill out a 30-minute questionnaire that includes questions on demographics (such as age, ethnicity, marital status, etc.), medication history, work history, hip surgeries, and assessment of functional disability. Fifty milliliters (about 3-1/3 tablespoons) of blood will be drawn for gene testing, and X-rays will be taken of the pelvis, lower back, and neck, if recent X-rays (within 1 year) are not available. Women of childbearing age will have a urine pregnancy test before having X-rays.

DETAILED DESCRIPTION:
The susceptibility to ankylosing spondylitis (AS) is largely genetically determined. Recent studies suggest that the severity of AS is also influenced to a large extent by genetic factors. The goal of this study is to identify genes that influence the severity of AS. We hypothesize that genetic markers of susceptibility, including human leukocyte antigen (HLA) polymorphisms, are among the genes that also influence the severity of AS. Other genes that could potentially influence the severity of AS include those that affect the severity of joint inflammation and those that influence bone formation.

In this cross-sectional study, we will test the association of HLA markers and polymorphisms in several genes involved in the regulation of inflammation and bone formation with the severity of AS. Approximately 500 patients will be enrolled. Each patient will have had AS for at least 20 years. Measures of AS severity will be the extent of spinal fusion as measured radiographically, functional disability, time to permanent work disability, and need for total hip arthroplasty.

Identifying genetic markers that are associated with differences in the severity of AS will greatly enhance our understanding of the pathogenesis of this disease by suggesting mechanisms and pathways involved in the development of long-term damage. In a separate but related protocol, we will assess genetic markers associated with persistent active inflammation in patients with AS.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Participants will:

1. have been diagnosed with AS by the modified New York criteria
2. have had AS for 20 years or more. The duration of AS will be dated from the time of onset of symptoms of inflammatory low back pain or restricted spinal motion
3. be able to read English.

Potential participants will be excluded if:

1. onset of AS was at age 16 or younger
2. have a spondyloarthropathy other than AS
3. are unable to provide informed consent.

Study of patients with AS for 20 years or more will provide a sample with a greater proportion of patients who will have developed the outcomes of interest. All participants will necessarily be age 37 or older. Study entry is not limited by sex or ethnic origin. English literacy is required because the functional status questionnaires used in the study have not been developed and validated in many languages other than English. In particular, the HAQ-S has been validated in only English, Dutch, and Finnish. The BASFI has been validated in English, Dutch, Finnish, Swedish, German, and French. Each of these validation studies consists of a single report. Monolingual speakers of these languages are likely to be rare in our area.

Potential participants will be recruited by physician referral and self-referral. Information about the study will be mailed to local rheumatologists and posted on the NIH website. Notices will also be sent to local chapters of the Arthritis Foundation and the Spondylitis Association of America.

Study of first-degree relatives:

Participants will be:

1. Parent, sibling, or child (age 18 or older) of an enrolled subject.
2. Able to provide informed consent.

Family members may by asymptomatic or have signs or symptoms of AS or a condition in the spondyloarthropathy family. There is no requirement for a minimum number of members per family to be eligible for participation.

The recruitment ceiling will be unlimited. Approximately 500 subjects will be recruited from all study sites. The target sample for the primary analyses will be 400 eligible subjects. Approximately 150 subjects will be recruited at the NIH.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2003-03-24 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Ward, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Gran JT, Skomsvoll JF. The outcome of ankylosing spondylitis: a study of 100 patients. Br J Rheumatol. 1997 Jul;36(7):766-71. doi: 10.1093/rheumatology/36.7.766. PMID 9255111
- [Background] Amor B, Santos RS, Nahal R, Listrat V, Dougados M. Predictive factors for the longterm outcome of spondyloarthropathies. J Rheumatol. 1994 Oct;21(10):1883-7. PMID 7837155
- [Background] Boyer GS, Templin DW, Bowler A, Lawrence RC, Everett DF, Heyse SP, Cornoni-Huntley J, Goring WP. A comparison of patients with spondyloarthropathy seen in specialty clinics with those identified in a communitywide epidemiologic study. Has the classic case misled us? Arch Intern Med. 1997 Oct 13;157(18):2111-7. PMID 9382668
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-AR-0130.html